CLINICAL TRIAL: NCT07161076
Title: Evaluation of a Novel 3D Printed Space Maintainer Versus the Conventional Stainless-Steel Band and Loop: A Finite Element Analysis and In-Vivo Study
Brief Title: Evaluation of a 3D Printed Space Maintainer Versus the Conventional Band and Loop
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Collaborators: Suez Canal University (Other)
Responsible Party: Principal Investigator, Omar hodhod, Assistant lecturer of pediatric dentistry, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 648/2023; 648/2023 (Other: Suez Canal University)
Record Dates: First submitted 2025-05-21; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Space Maintenance; 3D Printing; Primary Teeth
Keywords: 3d printing; resin 3d printed space maintainer; 3d printed; space maintainer; split mouth

STUDY DESIGN:
Intervention Model Description: Split Mouth
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metal Band and loop (Active Comparator): Classic Stainless-steel Band and Loop , Control group
  Interventions: Device: stainless steel band and loop
- 3d Printed Resin band and loop (Experimental): 3d printed band and loop with the new design , using Permanent Crown resin
  Interventions: Device: 3d Printed space maintainer

INTERVENTIONS:
Device: 3d Printed space maintainer — using Next dent permanent crown resin, a digitally designed space maintainer will be 3d printed to maintain space after extraction
  Arms: 3d Printed Resin band and loop
Device: stainless steel band and loop — lab fabricated metal band and loop
  Arms: Metal Band and loop

SUMMARY:
The goal of this study is to evaluate whether a new 3D-printed dental device can effectively maintain space after premature loss of primary teeth in children, compared to the traditional stainless-steel device. It will also assess safety and comfort. The main questions it aims to answer are:

1. What is the clinical success rate of 3D printed space maintainers compared to traditional metal band and loop space maintainers over a 12-month period?
2. How do 3D printed space maintainers compare in maintaining space and preventing rotation of abutment teeth?
3. What are the differences in gingival health outcomes between the two types of space maintainers?

Participants (13 children aged 6-9 years) will:

Receive both devices in a "split-mouth" design (one on each side of the mouth), totaling 26 treated tooth spaces (13 per group).

Attend checkups every 3 months for a year to monitor the devices' performance.

ELIGIBILITY:
Inclusion Criteria:

1. Apparently healthy children.
2. Children of both genders aged 6-9 years old.
3. Guardians agree to join the study and sign the informed consent.
4. Recent premature loss of primary first molars or having primary first molars indicated for extraction on both sides.
5. Sound buccal and lingual surfaces of abutment teeth (primary second molar and primary canine).
6. Good oral hygiene.
7. Absence of radiographic periapical pathology related to the abutment teeth.
8. Absence of abnormal occlusal conditions such as posterior crossbite, deep bite, and scissor bite.
9. All the indications for a band and loop space maintainer are met.

Exclusion Criteria:

1. The patient is not able to attend regular follow-up visits.
2. Allergic condition to any of the used materials.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 13 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Success Rate of Space Maintainers | 12 months
  Percentage of space maintainers remaining functional without failure
  Unit of Measure: Percentage of participants
Gingival health index | at 3-month follow-up, 6 months follow-up , and 1 year follow-up
  measuring Gingival index for both space maintainers to compare the a ability of plaque to attach to both devices. scale 0-3, higher scores indicate worse gingival health

SECONDARY OUTCOMES:
Wong-Baker FACES Pain Rating Scale | immediately after cementation,at 3-month follow-up
  Scale Range: 0 (no hurt) to 10 (hurts worst)
  Interpretation: Higher scores indicate worse pain/lower satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Omar A Hodhod, Principal Investigator — The British University in Egypt , Suez canal university
Locations (1):
- The British University in Egypt , Pediatric Dentistry Clinic, El Shorouk, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT07161076/Prot_SAP_ICF_000.pdf